CLINICAL TRIAL: NCT07051018
Title: Radiological and Clinical Measures as Predictors of Dynamic Postural Control Deficits in Chronic Ankle Instability
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Seif El-Eslam Youssif El-Said, Lecturer Assistant at faculty of physical therapy- University of Hertfordshire, Cairo University
Other Study IDs: P.T.REC/012/005628
Record Dates: First submitted 2025-04-06; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: postural control; chronic ankle instability; talar tilt; tibiotalar contact ratio

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to investigate the association between dynamic postural control and clinical measures of (ankle and hip strength, ankle DFROM and position sense) and radiological measures in patients with unilateral CAI.

DETAILED DESCRIPTION:
Ankle sprains are among the most frequent injuries seen in emergency departments and in sports injury clinics. Among all ankle injuries, ankle sprains are the most common and account for approximately 80% of which 77% are lateral sprains. Ankle sprain incidence ranges from 5.3- 7.0 sprained ankles per one thousand persons per year in Europe and is estimated to be 23,000 ankle sprains occur per day in the United States. Up to 74% of individuals who sprained their ankle experience ongoing problems that prevent them from participating in sports and other physical activities. Lateral ankle sprain (LAS) typically occurs when the rear foot is supinated, and the leg is externally rotated. Inversion injuries affect the lateral ankle ligaments and subtalar ligaments concomitantly; around 73% of lateral ankle sprains are due to rupture or tear of the Anterior Talo-Fibular Ligament (ATFL), followed by Calcaneo Fibular Ligament (CFL) and cervical ligament of the subtalar joint with the interosseous talocalcaneal ligament respectively.

HYPOTHESES:

It will be hypothesized that:

1. There will be no relation between the radiological measures of the ankle joint and dynamic postural control in patients with unilateral CAI.
2. There will be no relation between hip muscles strength and dynamic postural control in patients with unilateral CAI.
3. There will be no relation between ankle performance (muscle strength, DFROM and position sense) and dynamic postural control in patients with unilateral CAI.
4. There will be a non-significant difference in the dynamic postural control between affected and normal lower limb.
5. There will be a non-significant difference in the radiological measures between affected and normal lower limb.
6. There will be a non-significant difference in the ankle performance between affected and normal lower limb.
7. There will be a non-significant difference in the muscle strength around the hip joint between the affected and normal lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be screened for eligibility and only those who meet the inclusion criteria according to Delahunt et al. (2010) and Gribble et al. (2013) will be enrolled in our study, i.e., they will participate if they have:

  1. At least one significant unilateral lateral ankle sprain in which the subject was unable to walk independently without the aid of crutches (the first sprain occurred more than 12 months ago).
  2. Repeated bouts of lateral ankle injury (last injury had to be more than three months prior to inclusion in the study).
  3. Feeling of ankle instability "giving way", at least 2 episodes in the last 6 months (Terada et al., 2014).
  4. Pain during intense loading.
  5. The Cumberland Ankle Instability Tool (CAIT) ≤ 24.
  6. Age range of 18-30 years (Delahunt et al., 2010).

Exclusion Criteria:

* *Patients will be excluded if they didn't meet the inclusion criteria mentioned above, such as:

  1. A previous trauma or surgery to the trunk or lower extremities other than an ankle sprain.
  2. Neurological or vestibular impairments with remaining deficits.
  3. No participant with CAI had acutely sprained his or her ankle in the 3 months prior to the testing.
  4. Participants will be excluded if they have participated in any rehabilitation in the past 6 months.
  5. Concussion or head injury or lower back pain in the past 6 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 participants, with age between 18- 30 years, diagnosed with unilateral CAI will be recruited through direct referrals based on their availability to participate, thus, a sample of convenience will be used.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Y- balance test | baseline
  It is a dynamic balance test that assesses an individual's ability to maintain balance while reaching in three directions (anterior, posteromedial, and posterolateral) with one leg while standing on the other.

SECONDARY OUTCOMES:
Radiographic measurements validated for non weight bearing radiographs (Talocrural Angle and Talar Tilt) | baseline
  Tibiotalar contact ratio: this measurement represents congruency of the ankle joint on the lateral view . The measurements include the radius of the talus in mm, the height of the talus (h) in mm, and the tibiotalar sector (α) in degrees.
  Talar Tilt: It is the angle between the longitudinal axis of the tibia and joint orientation line of the tibiotalar joint. It is categorized as varus (< 87°), normal (87-91°) or valgus (> 91°) position of the ankle.

IPD SHARING:
Plan to Share IPD: Undecided